CLINICAL TRIAL: NCT00004145
Title: Allogeneic Peripheral Blood Stem Cell Transplantation Using a Non-Myeloablative Preparative Regimen for Patients With Hematologic Malignancies
Brief Title: Chemotherapy Plus Biological Therapy Followed By Peripheral Stem Cell Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9581; UCCRC-9581; UCCRC-CTRC-9852; NCI-G99-1618
Record Dates: First submitted 1999-12-10; First posted 2004-02-16 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Antilymphocyte Serum; Cyclophosphamide; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Fludarabine (30mg/m2/day x 5 days on days -9 to -5), cyclophosphamide (2gm/m2/day on day -5), antithymocyte globulin (10mg/kg/day x 4 days on days -5 to -2), tacrolimus (.03 mg/kg/day IVPB continuous infusion), mycophenolate mofetil (1mg PO BID, days +1 to +60), allogenic peripheral blood stem cells
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: fludarabine phosphate; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: cyclophosphamide
Drug: fludarabine phosphate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Sometimes the transplanted cells are rejected by the body's normal tissues. Antithymocyte globulin may prevent this from happening.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy plus biological therapy followed by peripheral stem cell transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of nonmyeloablative chemotherapy followed by allogeneic peripheral blood stem cell transplantation on hematopoietic recovery in patients with hematologic malignancies. II. Determine the toxicities of this regimen in these patients. III. Determine the frequency of mixed hematopoietic chimerism in these patients after this therapy. IV. Determine the efficacy and toxicity of donor leukocyte infusions at relapse in these patients. V. Determine the response rates and survival of these patients after this therapy. VI. Determine the immune reconstitution of patients undergoing this therapy.

OUTLINE: Patients receive fludarabine IV over 30 minutes on days -9 to -5, cyclophosphamide IV over 1 hour on day -5, and antithymocyte globulin IV over 10 hours on days -5 to -2. Allogeneic peripheral blood stem cells are infused on day 0. Patients who achieve complete remission (CR) and then relapse or patients who achieve less than a CR before day 60 receive donor leukocyte infusions (DLI) over 30 minutes. DLI are repeated as necessary for persistent disease. Patients are followed at 1, 3, and 6 months, then at 1 and 2 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven hematologic malignancy for which there is no standard curative therapy, including, but not limited to: Low grade non-Hodgkin's lymphoma (NHL) Mantle cell lymphoma Chronic lymphocytic leukemia (stage II-IV) Myelodysplastic syndrome, including: Refractory anemia (RA) with ringed sideroblasts RA with excess blasts (RAEB) RAEB in transformation Chronic myelomonocytic leukemia Multiple myeloma OR Histologically proven hematologic malignancy that has failed 1 prior therapy OR is at high risk for relapse, including, but not limited to: Intermediate grade NHL High grade NHL Hodgkin's disease Acute lymphoblastic lymphoma Acute myelogenous leukemia OR Histologically proven chronic myelogenous leukemia in chronic or accelerated phase, with the following risk factors that preclude eligibility for standard allogeneic peripheral blood stem cell transplantation: Older age Poor performance status Healthy, partially related HLA 5/6 or 6/6 serologic match donor available A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 to 60 or physiologic 70 Performance status: Karnofsky 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 2.0 mg/dL SGOT and SGPT less than 2 times normal No active hepatitis Renal: Creatinine less than 2.0 mg/dL OR Creatinine clearance greater than 50 mL/min Cardiovascular: Ejection fraction greater than 45% OR Cardiac clearance Pulmonary: DLCO at least 50% predicted Other: No active infection HIV-1, HIV-2, and HTLV-1 negative Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 1998-11; Primary Completion 2003-11 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Hematopoetic recovery and toxicities of non-myeloablative allogenic stem cell transplantation Hematopoetic recovery and toxicities of non-myeloablative allogenic stem cell transplantation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Zimmerman, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States